CLINICAL TRIAL: NCT03148743
Title: Department of Hematology of First Affiliated Hospital of Soochow University
Brief Title: FMT in Gut aGVHD Treated
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Qi Xiao-Fei, Principal Investigator, The First Affiliated Hospital of Soochow University
Other Study IDs: FMT2017002
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Acute-graft-versus-host Disease
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Fecal microbiota — fecal microbiota transplantation

SUMMARY:
With the stem cell transplanting increasing, patients which effected with gut GVHD were also increased. To evaluation the safety and efficacy of FMT for gut GVHD,patients with gut GVHD were recruited.

ELIGIBILITY:
Inclusion Criteria:

* gut GVHD

Exclusion Criteria:

* Age>60; or Age<10

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: After stem cell transplantating , some patients suffered the gut GVHD were recuited
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
times of stool | 24hours,48hours,72hours, 96hours,fifth day,sixth day, a week
  Change from stool times in a week

SECONDARY OUTCOMES:
volume in milliliter of stool | 24hours,48hours,72hours, 96hours,fifth day,sixth day, a week
  Change from stool volume in a week

CONTACTS AND LOCATIONS:
Overall Officials: depei wu, Study Chair — first affiliated of Soochow university
Locations (1):
- 中国, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Zhao Y, Qi J, Ma X, Qi X, Wu D, Xu Y. Fecal microbiota transplantation combined with ruxolitinib as a salvage treatment for intestinal steroid-refractory acute GVHD. Exp Hematol Oncol. 2022 Nov 9;11(1):96. doi: 10.1186/s40164-022-00350-6. PMID 36352455
- [Derived] Zhao Y, Li X, Zhou Y, Gao J, Jiao Y, Zhu B, Wu D, Qi X. Safety and Efficacy of Fecal Microbiota Transplantation for Grade IV Steroid Refractory GI-GvHD Patients: Interim Results From FMT2017002 Trial. Front Immunol. 2021 Jun 17;12:678476. doi: 10.3389/fimmu.2021.678476. eCollection 2021. PMID 34220825
- [Derived] Qi X, Li X, Zhao Y, Wu X, Chen F, Ma X, Zhang F, Wu D. Treating Steroid Refractory Intestinal Acute Graft-vs.-Host Disease With Fecal Microbiota Transplantation: A Pilot Study. Front Immunol. 2018 Sep 25;9:2195. doi: 10.3389/fimmu.2018.02195. eCollection 2018. PMID 30319644